CLINICAL TRIAL: NCT03301376
Title: INTHEMO: Occupational Integration of Adults With Severe Haemophilia in France: a Study Based on the FranceCoag Cohort
Brief Title: Occupational Integration of Adults With Severe Haemophilia in France: a Study Based on the FranceCoag Cohort
Acronym: INTHEMO
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-51
Record Dates: First submitted 2017-09-29; First posted 2017-10-04 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Severe Haemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Severe haemophilia and subsequent arthropathy result in joint pain, disability and impaired health-related quality of life. Improvements in haemophilia care over the last decades might lead to expectation of a near-normal quality of life for adults with haemophilia. However, little is known about the impact of haemophilia and its treatment on social functioning. A study based on a national US cohort of 141 young men (18-34 y.o.) showed that, compared to the general US population, this cohort experienced social burdens such as unemployment and lower high-school graduation rates. Another study conducted in the framework of the HERO (Haemophilia Experiences, Results and Opportunities) international initiative showed that a majority of the 230 young adults aged 18-30 years (including 16 French participants) were employed at least part-time (62%) and most of them reported that haemophilia has had a negative impact on employment (76%) which was reported as moderate or very large by 47% of the participants. The replicability of these results could be limited by the specific socio-economic national context. In France, a survey was conducted in 2008 to assess quality of life and its determinants in children, adolescents and adults with moderate and severe haemophilia. Descriptive results on the socio-economic characteristics of the included adults showed that 51.3% of them had access to higher education (which was higher than the observed rate in the French general population in 2005, i.e. 32.5%), and that 52.1% were employed among whom 44.3% had an at-risk activity. In spite of these results which were presented in a descriptive report by the InVS (Institut de veille sanitaire - French Institute for Public Health Surveillance), some limitations could be discussed:

DETAILED DESCRIPTION:
The principal objective of the present project is to assess occupational issues in an exhaustive national cohort of persons with severe haemophilia compared to the national population in order to describe the impact of severe haemophilia on the occupational integration.

Detailed objectives are mentioned hereinbelow:

1. To assess occupational issues in adults with severe haemophilia in France
2. To assess the impact of the changes of the context of life over the last decades in the new generation of adults with severe haemophilia in France
3. To compare occupational outcomes between adults with severe haemophilia and the general population in France
4. To identify individual characteristics (socio-demographics, clinical and psycho-behavioural) associated with occupational issues in adults with severe haemophilia in France
5. To compare occupational issues between adults with severe haemophilia and adults with others severe chronic childhood diseases in France to identify common and haemophilia-specific issues

Material and methods:

All adults (18-65 y.o.) participating in the FranceCoag cohort, which includes more than 1,500 French adults with severe haemophilia followed-up in 34 Haemophilia Treatment Centres, will be invited to participate in the study. These adults will be identified through the database of the FranceCoag cohort, and will be invited to participate through the post by the physician who follows them up in the Haemophilia Treatment Centre. If they agree to participate, they will be asked to fill a self-administered questionnaire in. This questionnaire will include items focusing on the following outcomes:

* occupational outcomes:

  * access to higher education and high-school graduation,
  * age at the start of working life,
  * degree of employment (unemployment / part-time employment / full-time employment),
  * sheltered employment,
  * job security (temporary / permanent contract / self-employment),
  * type of job (using the International Standard Classification of Occupations)
* socio-demographic outcomes:

  * age
  * living with a partner
  * having dependent children
* psycho-behavioural outcomes:

  * depressive symptomatology (using the Center for Epidemiologic Studies Depression (CES-D) scale)
  * quality of life (using the generic scale 36-Item Short Form Survey (SF-12) and the haemophilia-specific scale Haem-A-QoL)
  * anxiety (using the Strate-Trait Anxiety Inventory (STAI) scale)
  * coping strategies (using the BriefCOPE)
  * perceived impact of haemophilia on employment
  * participating in therapeutic education sessions
  * member of the Association française des hémophiles (AFH)

Clinical outcomes will be recorded via the FranceCoag cohort database (type of haemophilia, treatment, presence of an inhibitor, comorbidities as HIV and HCV infections).

Occupational outcomes of the participants will be described, and compared to the French national population. Expected distributions of the outcomes will be established by using data from the French National Institute for Statistics and Economic Studies. Observed and expected distributions will be compared. The modulating role of individual characteristics (including the period of birth, the presence of an inhibitor, comorbidities as HIV and HCV infections) in occupational issues will be assessed.

Expected results:

The results of this project will establish an updated picture of the occupational situation of French adults with severe haemophilia. By comparing the evolution of the occupational situation among them with the evolution in adults from the general population, the investigators will be able to assess the possibly different impact of the changes of the socio-economic context on the occupational situation of adults with severe haemophilia. The results will also establish a new picture of the occupational situation for the new generation of adults who was not concerned by the survey carried out about ten years ago. This sub-group is of particular interest as the impact of the disease on their life might have been different (major therapeutic progresses, no exposition to transfusion-transmitted infections).

Via the French haemophilia society (AFH) which is a partner of the present project, the results from the objectives 1 to 4 will be used for the education, training and awareness of patient resources, for the development of therapeutic patient education sessions focused on occupational issues, and for the drawing up of a brochure intended for patients.

Survivors of childhood leukemia from the French LEA cohort who present a higher rate of employment than the general population, but a lower access to a steady job could be an interesting comparative group for the fifth objective. As numerous actions are proposed to facilitate the occupational integration of survivors of cancer, the identification of the haemophilia-specific difficulties could help the decisions-makers to allocate means according to the specific needs of the persons with haemophilia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe haemophilia
* Patients aged from 18 to 65 years old
* Patients enrolled in the FranceCoag national cohort
* Patients affiliated to the French social security system
* Non opposition to participate in the study

Exclusion Criteria:

* Patients with moderate or minor haemophilia
* Patients under the age of 18 or over the age of 65
* Patients with comprehension problems
* Patients unable to read or to write
* Vulnerable patients
* Opposition to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults with severe haemophilia
Sampling Method: Non-Probability Sample
Enrollment: 590 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-05-27 (Actual)

PRIMARY OUTCOMES:
Degree of employment | one day
  unemployment / part-time employment / full-time employment

SECONDARY OUTCOMES:
Access to higher education and high-school graduation | one day
  Specific item of the patient questionnaire (yes(type)/no)
Age at the start of working life | one day
  Specific item of the patient questionnaire (age(years))
Sheltered employment | one day
  Specific item of the patient questionnaire (yes(type)/no)
Job security | one day
  Specific item of the patient questionnaire (temporary / permanent contract / self-employment)

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Hôpital de la Timone Assistance Publique Hôpitaux de Marseille, Marseille, France